CLINICAL TRIAL: NCT04458389
Title: Phase 1 (Dose Escalation)/Phase 2 (Expansion Cohort) Trial of TY101 as a Single Agent in Patients With Locally Advanced/Metastatic Solid Tumors and Relapsed or Refractory Lymphomas
Brief Title: A Phase 1/2 Study of TY101 for Locally Advanced /Metastatic Solid Tumors and Relapsed or Refractory Lymphomas
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tayu Huaxia Biotech Medical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TY101-001
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-05

CONDITIONS: Locally Advanced /Metastatic Solid Tumors; Relapsed or Refractory Lymphomas
MeSH Terms: conditions — Recurrence; Lymphoma

STUDY DESIGN:
Intervention Model Description: TY101 injection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TY101 (Experimental): Dose escalation：Humanized anti-PD-1 monoclonal antibody is to be injected intravenously 0.3mg/kg or 1mg/kg or 3mg/kg or 10mg/kg 200mg (fix dose) until disease progresses or unacceptable tolerability occurs.
  Dose expansion：After completion of the DLT observation, the sponsor and principal investigator will select a possible dose（RP2D）for dose expansion to further confirm the efficacy and safety of RP2D.
  Interventions: Drug: TY101

INTERVENTIONS:
Drug: TY101 — Dose escalation: TY101 0.3mg/kg or 1mg/kg or 3mg/kg or 10mg/kg 200mg Intravenous Q3W, 2 years depending on response.
  Dose expansion: Subjects received TY101 injection for a maximum of 2 years until progressive disease, intolerant toxicity, death, or withdrawal from the study occurred.

SUMMARY:
A multicenter, open-label, dose-escalation and dose-expansion phase 1/2 study, to evaluate TY101 safety, tolerability, pharmacokinetic characteristics, effectiveness and immunogenicity in patients with Locally Advanced /Metastatic Solid Tumors and Relapsed or Refractory Lymphomas. The study includes two parts: dose escalation and expansion cohort to evaluate the tolerability and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years
2. Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures.
3. Histological or cytological diagnosis, advanced solid tumor and lymphoma(Dose escalation phase), Or recurrence and refractory peripheral T-cell lymphoma who must have failure at least 1 prior routine regimen, or failure to tolerate the toxicity, or lack of any routine regimens, advanced squamous cell carcinoma of the skin and other advanced solid tumors and lymphoma (Dose expansion phase）
4. At least one evaluable lesion for solid tumor or lymphoma.
5. Must provide with tumor specimen that meet the requirements for biomarker testing(expression of PD-L1 and the infiltrating lymphocytes).
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at the screening and without deterioration within 2 weeks before enrollment.
7. Life expectancy ≥12 weeks
8. Adequate organ function as evidenced by meeting all the following requirements (with 14 days):

   1. Hemoglobin ≥ 9.0 g/dL neutrophils ≥ 1500 cells/ µL platelets ≥ 100× 10^3/ µL;
   2. Total bilirubin ≤ 1.5×upper limit of normal(ULN) aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5×ULN without, and ≤ 3×ULN with hepatic metastasis;
   3. International Normalized Ratio (INR) ≤1.5×ULN;
   4. Serum creatinine ≤1×ULN, creatinine clearance >60ml/min (Cockcroft-Gault equation).
9. The results of blood pregnancy tests must be negative for premenopausal women screened. All enrolled patients (male or female) should agree with adequate and reliable barrier contraception from signing informed consent date to the 6 months after the last dose.

Exclusion Criteria:

1. Previously received any of the following therapies:

   1.1 Received any other cytotoxic chemotherapeutic agents within 4 weeks prior to the first dose; for nitrosoureas and mitomycin C at least 6 weeks.

   1.2 Received any targeted or other anticancer drug therapy within 4 weeks prior to the first dose.

   1.3 Radiation therapy within 4 weeks prior to first dose (note: palliative radiotherapy for bone or palliative radiotherapy for superficial lesions was allowed, the course of treatment is based on local standards and had been ended 2 weeks before the first dose. Radiotherapy covering more than 30% of the bone marrow area within 4 weeks prior to first dose was excluded).

   1.4 NMPA-approved antitumor Chinese traditional medicine is in use or has been used within 2 weeks prior to the first dose.
2. Concurrent malignancy within 5 years prior to screening, except for the cured basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
3. Patients with active central nervous system (CNS) metastasis and/or cancerous meningitis who were found on known or in the screening tests, except for the following subjects: Subjects with asymptomatic brain metastasis who need to undergo regular brain imaging examination as the site of the disease. Subjects with stable status of brain metastasis after treatment.
4. Concomitant active or suspected autoimmune disease; but patients who are in a stable state and did not require systemic immunosuppressive therapy are allowed to be enrolled.
5. A history of allogeneic organ, bone marrow transplant or stem cell transplant; A history of allogeneic organ, bone marrow or stem cell transplantation.
6. Patients with the history of or are suffering from pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe pulmonary function impairment, etc., which may interfere with the detection and management of suspected drug-related pulmonary toxicity; patients with active tuberculosis or with a history of active tuberculosis infection ≤48 weeks prior to screening, regardless of treatment.
7. Severe cardiovascular disease, such as NYHA class III or IV congestive heart failure. A history of myocardial infarction, poorly controlled arrhythmias (including QTc interphase ≥450 ms in men and ≥470 ms in women, as calculated by the Fridericia formula), or cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis, and pulmonary embolism in the 6 months prior to screening.
8. Uncontrolled hypertension (systolic blood pressure >150 mmHg and diastolic blood pressure > 100 mmHg), a history of hypertension crisis, or a history of hypertensive encephalopathy.
9. Uncontrolled endocrine diseases (diabetes, thyroid disease, etc.).
10. Patients with active peptic ulcer or hemorrhagic disease.
11. Seriously infected persons who need to be treated with systemic antiviral or antimicrobial treatment.
12. Pericardial effusion, pleural effusion and peritoneal effusion that remained uncontrolled after intervention.
13. Patients with any other severe, acute or chronic disease that the investigator considers to be likely to interfere with participation in the study or evaluation and which the investigator determines to be inappropriate for participation in the clinical trial.
14. HIV infection.
15. Active viral hepatitis patients are excluded. Patients with serologic evidence of chronic HBV infection (defined by a positive hepatitis B surface antigen test and a positive anti-hepatitis core antigen antibody test, and the HBV-DNA); HCV infection (defined by positive HCV antibody and HCV-RNA test).
16. The history of other therapies against immune checkpoint, such as anti-PD-1, anti-PD-L1, anti-CTLA-4 or anti-LAG-3.
17. Have received steroids or other systemic immunosuppressive therapy within 14 days prior to the first dose, or have to be treated while on trial; except the following: a) The use of topical or inhaled corticosteroids, b) Glucocorticoids are used in the short term (continuous use≤7 days) to prevent or treat non-autoimmune allergic diseases.
18. History of serious allergic reaction to treatment with another monoclonal antibody.
19. A history of alcohol, drug or substance abuse.
20. Major surgery within 4 weeks prior to screening or scheduled to undergo major surgery during the trial.
21. Live virus vaccine or attenuated vaccine within 30 days prior to first dose.
22. Be in the other clinical studies now, or have participated in other intervention clinical trials in the previous 4 weeks.
23. Pregnant or breast-feeding females.
24. Any condition that the investigator believes may not be appropriate for participating the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability measured | 90 days after the last dose.
  Number of Participants with treatment-related Adverse Events (AEs) by CTCAE v5.0.
Dose-limiting toxicity(DLT) | 3 weeks after first dose for each dose group.
  DLT is the primary endpoint for safety in the dose escalation phase and will be used to determine the maximum tolerated dose (MTD).

SECONDARY OUTCOMES:
Pharmacokinetics(Cmax) | Up to approximately 12 months
  Maximum Concentration(Cmax)
Pharmacokinetics(Tmax) | Up to approximately 12 months
  Dose escalation: Peak time(Tmax)
Pharmacokinetics(AUC) | Up to approximately 12 months
  Dose escalation: Area Under Curve(AUC)
Pharmacokinetics(t1/2) | Up to approximately 12 months
  Dose escalation: half life(t1/2)
Pharmacokinetics(PPK) | The PPK evaluation will be further designed based on the results of the dose escalation phase.
  Dose escalation: Population pharmacokinetics(PPK)
Objective response rate(ORR) | Up to approximately 12 months
  Efficacy observation
Overall Survival(OS) | Up to approximately 12 months
  Efficacy observation
Progression-free survival(PFS) | Up to approximately 12 months
  Efficacy observation

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided